CLINICAL TRIAL: NCT04948918
Title: Efficacy of Distal Renal Denervation for Preventing Decline in Renal Function in Patients With Type 2 Diabetes Mellitus and Hypertension
Brief Title: Distal Renal Denervation to Prevent Renal Function Decline in Patients With T2DM and Hypertension
Acronym: REFRAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 005/e3
Record Dates: First submitted 2021-06-24; First posted 2021-07-02 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Type 2 Diabetes Mellitus; Hypertension
Keywords: hypertension; diabetes mellitus; kidney; renal function; denervation; blood pressure
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Distal renal denervation (Experimental): The arm comprises patients undergoing distal bilateral radiofrequency renal denervation performed using Symplicity Spyral renal denervation system.
  Interventions: Procedure: Anatomically optimized distal renal denervation

INTERVENTIONS:
Procedure: Anatomically optimized distal renal denervation — Bilateral radiofrequency renal denervation will be performed using Symplicity Spyral renal denervation system. Generally, at least two separate applications of radiofrequency energy will be performed in each segmental branch of renal artery. Each application will be done through 4 electrodes deployed in helical manner according to the design of the catheter

SUMMARY:
The aim of this study is to test the hypothesis that distal renal denervation (RDN) may delay or prevent the progressive decline of renal function in patients with type 2 diabetes mellitus and hypertension

DETAILED DESCRIPTION:
Detailed Description: Diabetes mellitus and hypertension are two major causes of chronic kidney disease (CKD) that starts as subclinical decline in renal function that silently progresses to symptomatic advanced stages associated with irreversible significant damage of the kidney structure. Recent major improvements in pharmacotherapy of hypertension and diabetes have substantially reduced the prevalence of cardiovascular complications, yet, the frequency of CKD remains largely unchanged. Renal denervation is a new minimally invasive method to create regional blockade of the renal sympathetic nerves that is currently used as non-pharmacological therapy of hypertension. The CKD is likewise mediated by overactivity of renal sympathetic system so that RDN has strong potential to prevent development or progression of CKD. The new anatomically optimized distal RDN may have additional benefit in this regard. Denervation of the distal vessels involved in tonic regulation of renal blood should cause a significant drop in renal vascular resistance and proportional increase in blood and oxygen supply to the kidney preventing/reducing chronic hypoxia of renal tissue that is major mechanism of CKD. The aim of this study is to prove the aforementioned concept. For this purpose the eligible patients with type 2 diabetes mellitus and hypertension will undergo distal renal denervation performed using dedicated radiofrequency catheter Symplicity Spyral. The changes in the kidney function and structure as well as BPs (office and ambulatory) will be assessed at baseline, 6 and 12 months post-procedure

ELIGIBILITY:
Inclusion Criteria:

* informed consent of participation in the study;
* systolic BP > 140 or diastolic BP > 90 mm Hg;
* type 2 diabetes mellitus (glucose tolerance test > 11.0 mmol/l, HbA1c>6,5%);

Exclusion Criteria:

* secondary hypertension;
* type 1 diabetes mellitus;
* acute renal failure;
* traumatic kidney injury;
* toxic kidney injury;
* CKD G4 and G5 according to the KDIGO 2012;
* infectious diseases requiring active antibacterial and/or antiviral therapy;
* other severe diseases and conditions

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Change in estimated glomerular filtration rate renal function (eGFR) | from baseline to 12 months
  eGFR calculated using CKD-EPI formula

SECONDARY OUTCOMES:
Change in eGFR | from baseline 12 months
  eGFR calculated using CKD-EPI formula
Change in office blood pressure levels (systolic/diastolic) | from baseline to 6 months and 12 months
  Blood pressure measurement performed by physician in office
Change in ambulatory 24-hour blood pressure levels (24-h mean, daytime, nighttime; systolic/diastolic) | from baseline to 6 and 12 months
  Mean values for respective periods calculated from ambulatory blood pressure monitoring performed using automatic measurement device
Change in cystatin C levels | from baseline to 6 and 12 months
  blood analysis
Change in lipocalin 2 (NGAL) levels | from baseline to 6 and 12 months
  blood analysis
Change in 24-hour urinary albumin excretion | from baseline to 6 and 12 months
  urinalysis
Change in the cortical and medullary volume of the kidneys and their ratio according to MRI | from baseline to 12 months
  Cortical and medullary volume measured using magnetic resonance imaging
Prognostic significance of baseline HbA1c value with regard to change in eGFR | from baseline to 6 and 12 months
  Will be assessed from multiple regression model of linear dependence of change in eGFR on a number of independent variables including in addition to HbA1c also age, sex, baseline eGFR, and 24-h ambulatory systolic BP
Change in renal resistive index in a trunk | from baseline to 6 and 12 months
  resistive index calculated using blood flow velocity on Doppler ultrasound
Change in peak linear blood flow velocity in the trunk and in segmental renal arteries | from baseline to 6 and 12 months
  blood flow velocity assessed by Doppler flowmetry in the trunk of the renal arteries and in segmental renal arteries using averaged values

CONTACTS AND LOCATIONS:
Overall Officials: Alla Falkovskaya, MD, PhD, Study Director — Cardiology Research Institute, Tomsk National Research Medical Centre, Russian Academy of Sciences
Locations (1):
- Cardiology Research Institute, Tomsk National Research Medical Centre, Russian Academy of Sciences, Tomsk, Russia